CLINICAL TRIAL: NCT06130267
Title: The Impact of an Immersive Digital Therapeutic Tool on Pain Perception: An Experimental Study With an Active Control Condition
Brief Title: The Impact of an Immersive Digital Therapeutic Tool on Pain Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stéphane Potvin (Other)
Responsible Party: Sponsor-Investigator, Stéphane Potvin, Full-time professor, Ciusss de L'Est de l'Île de Montréal
Organization: Ciusss de L'Est de l'Île de Montréal (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2022-2849
Record Dates: First submitted 2023-11-05; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Pain Perception
Keywords: Pain; Emotions; virtual reality; within-subject design
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control condition (Placebo Comparator): same paradigm without the active agent
  Interventions: Other: Endocare
- Virtual Reality condition (Experimental): calming VR environment
  Interventions: Other: Endocare

INTERVENTIONS:
Other: Endocare — Virtual paradigm (calming environnement)

SUMMARY:
The goal of this experimental study is to examine the impact of a virtual reality paradigm on heat pain perception in healthy volunteers. The main question it aims to answer is to determine if the virtual reality paradigm reduces pain intensity and unpleasantness evoked by tonic heat pain stimulation. Tonic heat pain stimulation is applied on the left forearm of participants using a Peltier thermode immediately before, during and immediately after virtual reality exposure. Using a with-subject design, participants are sequentially exposed to both the virtual reality condition and an active control condition. The order of administration of the virtual reality and control conditions is randomized.

DETAILED DESCRIPTION:
Pain is a complex and multifaced sensory and emotional experience. Virtual reality has shown promise in reducing experimental pain and chronic pain. However, many previous trials in the field lacked proper control conditions. This experimental study examines an immersive virtual environment initially designed for the treatment of endometriosis patients, which demonstrated promising analgesic effects. The current study aims to determine the impact of the virtual reality paradigm on experimental pain perception both during and after virtual reality exposure, while using an active control condition. This study involves healthy individuals with no chronic pain and uses a within-subject design, comparing a virtual reality paradigm with an active control condition. Continuous heat pain stimulation is applied to the left forearm of participants with a Peltier thermode, before, during and immediately after virtual reality exposure. For each continuous heat pain stimulation, pain intensity and unpleasantness are measured using a scale from 0 (no pain) to 100 (worst pain). Using a with-subject design, participants are sequentially exposed to both the virtual reality condition and an active control condition. The order of administration of the virtual reality and control conditions is randomized. Both conditions are administered in a single experimental session at the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* between 18 and 50 years old
* willing to participate in the study
* able to sign the informed consent form

Exclusion Criteria:

* neurological disorders
* substance use disorders
* severe mental health disorder
* chronic pain
* any acute and unstable medical condition
* taking medication that acts on the central nervous system

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Thermal heat pain induced with a Peltier thermode | Immediately before, during and immediately after VR exposure
  Pain intensity and unpleasantness, on a COVAS scale from 0 (no pain) to 100 (worse pain)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Potvin, PhD, Study Director — University of Montreal, Centre de recherche de l'institut universitaire en santé mentale de montréal
Locations (1):
- Centre de recherche de l'institut universitaire de santé mentale de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Diallo S, Marchand S, Dumais A, Potvin S. The impact of an immersive digital therapeutic tool on experimental pain: a pilot randomized within-subject experiment with an active control condition. Front Pain Res (Lausanne). 2024 Jun 6;5:1366892. doi: 10.3389/fpain.2024.1366892. eCollection 2024. PMID 38903416